CLINICAL TRIAL: NCT04697745
Title: Comparison Between Analgesic Effect of Dexamethasone and Dexmedetomidine as an Adjuvant to Bupivacaine for Spinal Anesthesia for Elective Caesarean Sections
Brief Title: Dexamethasone and Dexmedetomidine as an Adjuvant to Spinal Anesthesia for Elective Caesarean Sections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Baher Said Elshahat Mohamed Abdelhady, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: adjuvant to spinal anesthesia
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone intrathecal (Active Comparator)
  Interventions: Drug: Intrathecal dexamethasone
- dexmedetomidine intrathecal (Active Comparator)
  Interventions: Drug: Intrathecal dexmedetomidine

INTERVENTIONS:
Drug: Intrathecal dexamethasone — intrathecal adjuvants to bupivacaine
  Arms: dexamethasone intrathecal
Drug: Intrathecal dexmedetomidine — intrathecal adjuvants to bupivacaine
  Arms: dexmedetomidine intrathecal

SUMMARY:
The main objective of our study is to evaluate analgesic effect of intrathecal dexamethasone and dexmedetomidine in elective caesarean sections

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classII-III adult female patient (age :18 -40 years old )
* Elective cesarean section under spinal anaesthesia
* Gestational age > 37 weeks
* BMI less than 30 kg/m2

Exclusion Criteria:

* Patient refusal
* unable to give consent
* age < 18 or > 40
* BMI more than 30 kg/m2
* known allergy to the study medication
* coagulopathies or on anticoagulant medications
* diabetic neuropathy
* patients with psychiatric disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
analgesic effect | Up to 24 hours after surgery
  Duration of sensory block and time to first analgesic rescue .
  .

SECONDARY OUTCOMES:
intraoperative complications | during surgery
  Incidince of intraoperative shivering, nausea and vometing